CLINICAL TRIAL: NCT03788122
Title: Qualitative In-depth Interviews With Women and Their Partners Concerning the Acceptability of Fetal Surgery
Brief Title: Fetal Surgery Interview Study: Parental Perceptions of Fetal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University College, London (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S61586
Record Dates: First submitted 2018-12-13; First posted 2018-12-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Fetal Surgery; Myelomeningocele; Congenital Diaphragmatic Hernia
Keywords: Acceptability; Qualitative research; Patient Perspectives
MeSH Terms: conditions — Meningomyelocele; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents eligible for fetal surgery (Other): Parents eligible for fetal surgery will undergo two or three in-depth face-tot-face interviews, to determine their perception of acceptability of fetal surgery.
  Interventions: Other: In-depth interview

INTERVENTIONS:
Other: In-depth interview — The 'intervention' administered to this group of participants are two or three in-depth interviews (average 30-60 m minutes per interview) on their experiences, views, feelings and thoughts (perceptions) regarding acceptability of the fetal surgery.

SUMMARY:
Open maternal-fetal surgery is currently used on fetuses with myelomeningocele (MMC). Fetoscopic or minimal access fetal surgery is also being used to treat fetuses with congenital diaphragmatic hernia (CDH).

Following accurate diagnosis of a congenital malformation such as MMC or CDH, prospective parents face a range of uncertainties regarding the future of their unborn child, and the options provided require major ethical considerations. In the situation under study, termination of pregnancy may be for some parents an alternative option to expectant prenatal management. Fetal therapy provides a tantalising third option for some, where procedures are undertaken to reduce the likelihood of a more complicated neonatal course, potentially improving long term outcome, but at risk of amniotic fluid leakage, infection and most importantly very preterm delivery, itself associated with significant neonatal mortality and morbidity and long-term consequences. Balancing these competing risks is challenging.

For an intervention to be effective it also needs to be acceptable to women and their families. "Acceptability" can be defined as a multi-faceted construct that reflects the extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention.

With this study it is the aim to assess how women (and their partners) perceive the acceptability of a fetal surgical intervention for MMC and CDH. Participants will be asked to share their thoughts, views, feelings and experiences with regards to the decision to participate in fetal surgery. Data are collected by the use of in-depth face-to-face interviews. In-depth interviews are used to understand the participant's perspectives and perceptions of a situation they are in. It explicitly includes participants interpretation and understanding of an event

The interviews will be held in two or three moments in time (for parents opting for fetal surgery, there will be one additional interview, after the intervention while admitted in hospital): after counselling for options, but before eventual intervention; for intervention group shortly after the intervention, and 12 weeks after birth of the baby, or termination of pregnancy.

DETAILED DESCRIPTION:
1. Background and rationale Fetal surgery is a highly technical procedure carried out by only a few specialised teams around the world. Fetal surgery improves outcomes for key conditions, but at significant procedure related fetal and maternal risk. Open maternal-fetal surgery is currently used on fetuses with myelomeningocele (MMC). Fetoscopic or minimal access fetal surgery is also being used to treat fetuses with congenital diaphragmatic hernia (CDH). By combining improved instrumentation, imaging, clinical training and public engagement The Guided Instrumentation for Fetal Therapy and Surgery (GIFT-Surg) project aims to provide fetal surgeons with tools to make fetal surgery safer and more efficient. The UZ and KU Leuven team participates in this engineering project.

   Following accurate diagnosis of a congenital malformation such as MMC or CDH, prospective parents face a range of uncertainties regarding the future of their unborn child, and the options provided require major ethical considerations. In the situation under study, termination of pregnancy may be for some parents an alternative option to expectant prenatal management. Fetal therapy provides a tantalising third option for some, where procedures are undertaken to reduce the likelihood of a more complicated neonatal course, potentially improving long term outcome, but at risk of amniotic fluid leakage, infection and most importantly very preterm delivery, associated with significant neonatal mortality and morbidity and long-term consequences. Balancing these competing risks is challenging.
   1. Myelomeningocele Prevalence, incidence, clinical presentation Myelomeningocele (MMC) or spina bifida is a congenital abnormality arising 28 days post-conception when part of the neural tube fails to close. Open spina bifida can present either with a flat defect without a fluid filled sac covering (myeloschisis), or membranous covering with extrusion of the cord into the sac (myelomeningocele). Its prevalence is approximately 4.9 per 10,000 live births in Europe. Myelomeningocele is a severe, yet non-lethal congenital abnormality affecting the central nervous system, with complex physical and neurodevelopmental sequelae. In most cases it is also associated with the Chiari Type II malformation (hindbrain herniation) and ventriculomegaly.

      Therapy, risks and (long-term) outcome Until recently, the only options available to parents, once a diagnosis was made prenatally, were expectant management with delivery and postnatal surgery, or a pregnancy termination. But over the last thirty years, it became obvious that the condition is progressive in utero, as is suggested by the "two-hit" hypothesis; an initial embryonic failure in neurulation followed by secondary changes because of continuous exposure of the spinal cord to the intrauterine environment and the suction gradient on the hindbrain. This led to the concept of fetal intervention to arrest or reverse this natural course. Successful fetal coverage of MMC with improved functional outcome in the lamb model was first described in the late 1990s. This was translated clinically with encouraging early results in several case series and eventually led to the randomized controlled Management of Myelomeningocele Study (MOMS). This study demonstrated that mid-gestational layered repair reduces the need for ventriculoperitoneal shunting, improves the degree of hindbrain herniation, and preserves motor function better than postnatal surgery. However, fetal surgery for spina bifida comes with substantial maternal and fetal risks. The fetus is at increased risk of premature birth and its sequelae including sepsis, intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis and death. Besides there is the risk for maternal complications and the corporeal scar compromises uterine integrity.
   2. Congenital diaphragmatic hernia Prevalence, incidence, clinical presentation Due to a defect in the diaphragm during embryonic development, abdominal organs herniate through the defect into the thoracic cavity, interfering with lung growth, resulting in developmental arrest of both airways and pulmonary vasculature. Congenital diaphragmatic hernia (CDH) occurs in 1/2500 to 1/5000 births, depending on whether stillbirths are included. Although the diaphragmatic defect is correctable after birth, the prenatal arrest of airway and vessel development is the main reason for postnatal problems, leading to respiratory failure and pulmonary hypertension (PHT) in the neonatal period. Although prenatal referral to specialist centers, high throughput and advanced neonatal care has improved survival, still 20-30% of all cases die. Besides, survivors experience ongoing pulmonary and nutritional morbidity.

      Therapy, risks and (long-term) outcome In fetuses with poor prognosis, fetal lung growth can be stimulated by fetoscopic endoluminal tracheal occlusion (FETO) with a balloon. The fetal lung is a net secretor of fluid into the amniotic cavity and the lungs are maintained at a small positive pressure in normal development. Fetal tracheal occlusion (TO) prevents egress of lung liquid, leading to increased back pressure, in turn promoting stretch-induced growth of airways and vessels. TO appears to trigger sufficient lung growth to protect the lung from developing pulmonary hypoplasia. In utero reversal of the occlusion prompts pulmonary maturation. Experimentally an endoscopic technique of tracheal occlusion using a balloon was developed. In 2004, it was first applied clinically and referred to as Fetoscopic Endoluminal Tracheal Occlusion (FETO).

      The major risk following the procedure is spontaneous pre-labour rupture of membranes before 37 weeks (PPROM). Gestational age at delivery logically is an important predictor of survival and morbidity in CDH fetuses, also when undergoing fetal therapy.

      A meta-analysis suggests that FETO improves survival, but the procedure remains to be considered investigational and is therefore currently evaluated within a randomized controlled clinical trial (www.totaltrial.eu).
   3. Acceptability For an intervention to be effective it also needs to be acceptable to women and their families. "Acceptability" can be defined as a multi-faceted construct that reflects the extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention. Based on this definition a theoretical framework of acceptability comprising seven components has been developed: affective attitude, burden, perceived effectiveness, ethicality, intervention coherence, opportunity costs, and self-efficacy. Successful implementation of an intervention means that it is acceptable for both recipients and deliverers. This study focuses on the recipients; measurement of acceptability for deliverers will be considered as other facets of the wider GIFT-Surg project.

   Timing is an important factor in the assessment as the relationship to perceived and actual experiences may differ. Acceptability is therefore assessed in two or three moments in time: prospective acceptability, concurrent acceptability and retrospective acceptability.
2. Trial objectives

   Primary objective: to assess how women (and their partners) perceive the acceptability of a fetal surgical intervention for MMC and CDH. Participants will be asked to share their thoughts, views, feelings and experiences with regards to the decision to participate in fetal surgery.
3. Trial Design

   This is a qualitative in-depth interview study, to include approximately 48 women/couples at University Hospital Leuven for two fetal conditions (MMC and CDH), given all data on these 48 patients are complete. An estimated dropout rate of 50% means that in total 4 patients per treatment option (fetal surgery, expectant management, termination), and per condition (MMC or CDH) will be available for analysis.

   As not all parents opt for fetal surgery, after referral and counselling for prenatal diagnosed isolated spinal defects and congenital diaphragmatic hernia, patients fall into three groups: 1. Parents opting for fetal surgery, 2. Parents opting for termination of pregnancy and 3. Parents opting for expectant management. To assess acceptability of the intervention, it is of value to assess acceptability of the intervention in all three groups. In particular, knowledge of non-acceptability important.
4. Trial Intervention

   Data collection will take place by executing face-to-face interviews. The interviews will be held in three moments in time: before, during (i.e. shortly after the intervention) and after the intervention. Prospective acceptability will be assessed, after patients have been first counselled and assessed, but before the intervention at stake. Concurrent acceptability, patients will be interviewed shortly after the intervention while still admitted for post-surgery observation, and retrospective acceptability three months after delivery.

   The interviews assessing prospective and concurrent acceptability will always be planned along visits to the treatment hospital so parents never have to come on purpose to the hospital for an interview, and will be held in Dutch or English. The interviews are expected to last approximately 30-60 minutes and will follow an interview guide. As it is acknowledged women (and their partners) go through an intensive and emotionally upsetting process, interviews will only be carried out if the patient is capable of participating in an interview, based on the patient's personal assessment as well as their doctor's assessment. For retrospective acceptability, depending on participant's preference, the interview can take place through teleconference or phone.

   Data-collection Data are collected by the use of in-depth interviews. In-depth interviews are used to understand the participant's perspectives and perceptions of a situation they are in. It explicitly includes participants interpretation and understanding of an event. The style of interviewing will be 'responsive'; this style emphasises on the importance of building a relationship of trust between interviewer and interviewee. This is done by creating a quiet and calm environment, an empathically neutral position of the interviewer and an open approach by using verbal and non-verbal communication. There will not be a set list of questions, but an interview guide based on one main-question, with different themes for probing, based on the seven components of the framework of acceptability. The interview will follow six stages as described by Yeo et al.: arrival and introduction: establish rapport, 'host' the interaction(stage 1); introducing the research (aims and objectives, confidentiality, voluntary, scope of interview (participant in control), no right or wrong answers(stage 2); beginning of the interview: discuss contextual background information for reference and set the tone (stage 3); during the interview (start recording: breadth and depth of subject)(stage 4); ending the interview: advance notice of end and opportunity for respondent to raise anything important not yet discussed (stage 5); and after the interview: thanking and emphasize on value of sharing their experience, how information is treated and used, follow up and further meetings to be scheduled (stage 6)(interview guide).

   The interviews will be recorded digitally with an audio recorder. Subsequently, interviews will be transcribed and coded transcripts will be translated into English and used for analysis. Back-translation will be used for a sample of 5 transcripts in Dutch to ensure accuracy.
5. Sample size

   Intended sample size in Belgium is 12 women for MMC and 12 for CDH at study completion; in the UK the investigators expect to include 10 women for MMC and 5 for CDH. This sample size has been determined from interviewing clinical stakeholders. Sample size in qualitative research are usually small, as in analysis there will be at some point a moment in which no new information is obtained from additional interviews. This is also called saturation. The aim of this research is not to determine statistically significant discriminatory variables, but to get an in-depth understanding of the views and preferences of the participants, and to assess acceptability of the intervention. Exact sample size will depend on saturation
6. Analysis

The analysis is purely qualitative. The interviews will be transcribed verbatim by the researcher. Content analyses will be performed by using the qualitative software programme. First, initial content and subjects of interest are identified, the so-called familiarization with the data. This first step is followed by the initial construct of a framework. The framework constructs the headings under which respondent's views, feelings, experiences and perceptions can be organized. The framework is than used for labelling the data: quotes or pieces of text are ordered according to the different themes to fit in. The next step will be further refinement of the framework by making connections between categories and placing them in a broader context related to the framework of acceptability. To improve the quality of the analysis, at various moments interim analyses will be discussed among co-authors with a background in psychology and qualitative analysis. Thereafter, all previously analyzed transcripts will be reviewed to check that the content is consistent with this concept (thematic analysis).

ELIGIBILITY:
Inclusion Criteria:

* Women/partners eligible for one of the two fetal surgery procedures studied (open fetal surgery for spina bifida closure, tracheal balloon occlusion for congenital diaphragmatic hernia (Fetoscopic Endoluminal Tracheal Occlusion, FETO), as clinical care
* Have given written informed consent for participation

Exclusion:

* Women less than 18 years or over 65 years of age
* Partners less than 18 years or over 65 years of age
* Women or their partners who are unable to communicate in either English or the local language (if different)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Prospective acceptability of fetal surgery in the context of Myelomeningocele and Congenital Diaphragmatic Hernia. | After evaluation and counseling, if applicable, before undergoing fetal surgery.
  Qualitative methodology. Prospective acceptability, as perceived by prospective parents eligible for fetal surgery, assessed by in-depth face-to face interviews.
Concurrent acceptability of fetal surgery in the context of Myelomeningocele and Congenital Diaphragmatic Hernia. | After fetal surgery, within 7 days after surgery.
  Qualitative methodology. Concurrent acceptability, as perceived by prospective parents eligible for fetal surgery, assessed by in-depth face-to face interviews.
Retrospective acceptability of fetal surgery in the context of Myelomeningocele and Congenital Diaphragmatic Hernia. | Three months after birth of the baby, or three months after termination of the pregnancy.
  Qualitative methodology. Retrospective acceptability, as perceived by prospective parents eligible for fetal surgery, assessed by in-depth face-to face interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Deprest, Professor, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Neil Marlow, Principal Investigator — University College London Hospital
Locations (2):
- University Hospital Leuven, Leuven, Belgium
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen AR, Couto J, Cummings JJ, Johnson A, Joseph G, Kaufman BA, Litman RS, Menard MK, Moldenhauer JS, Pringle KC, Schwartz MZ, Walker WO Jr, Warf BC, Wax JR; MMC Maternal-Fetal Management Task Force. Position statement on fetal myelomeningocele repair. Am J Obstet Gynecol. 2014 Feb;210(2):107-11. doi: 10.1016/j.ajog.2013.09.016. Epub 2013 Sep 18. PMID 24055581
- [Background] Deprest J, Nicolaides K, Done' E, Lewi P, Barki G, Largen E, DeKoninck P, Sandaite I, Ville Y, Benachi A, Jani J, Amat-Roldan I, Gratacos E. Technical aspects of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia. J Pediatr Surg. 2011 Jan;46(1):22-32. doi: 10.1016/j.jpedsurg.2010.10.008. PMID 21238635
- [Background] Ville Y. Fetal therapy: practical ethical considerations. Prenat Diagn. 2011 Jul;31(7):621-7. doi: 10.1002/pd.2808. Epub 2011 Jun 10. PMID 21660998
- [Background] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- [Background] Al-Maary J, Eastwood MP, Russo FM, Deprest JA, Keijzer R. Fetal Tracheal Occlusion for Severe Pulmonary Hypoplasia in Isolated Congenital Diaphragmatic Hernia: A Systematic Review and Meta-analysis of Survival. Ann Surg. 2016 Dec;264(6):929-933. doi: 10.1097/SLA.0000000000001675. PMID 26910202
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Farmer DL, Thom EA, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Gupta N, Adzick NS; Management of Myelomeningocele Study Investigators. The Management of Myelomeningocele Study: full cohort 30-month pediatric outcomes. Am J Obstet Gynecol. 2018 Feb;218(2):256.e1-256.e13. doi: 10.1016/j.ajog.2017.12.001. Epub 2017 Dec 12. PMID 29246577
- [Background] Johnson MP, Bennett KA, Rand L, Burrows PK, Thom EA, Howell LJ, Farrell JA, Dabrowiak ME, Brock JW 3rd, Farmer DL, Adzick NS; Management of Myelomeningocele Study Investigators. The Management of Myelomeningocele Study: obstetrical outcomes and risk factors for obstetrical complications following prenatal surgery. Am J Obstet Gynecol. 2016 Dec;215(6):778.e1-778.e9. doi: 10.1016/j.ajog.2016.07.052. Epub 2016 Aug 2. PMID 27496687